CLINICAL TRIAL: NCT03516513
Title: Participatory Design of Electronic Health Record Tools for Problem Solving Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ian Bennett, Professor, School of Medicine: Family Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00004274; 1P50MH115837-01 (NIH)
Record Dates: First submitted 2018-03-28; First posted 2018-05-04 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Phase 1 will consist of qualitative interviews; Phase 2 will consist of rapid iterative design that includes qualitative interviews; Phase 3 will be an interventional pilot randomized trial. Data reported on ClinicalTrials.gov are for Phase 3.
Who Masked: Outcomes Assessor
Masking Description: Research Assistants and expert raters will not be informed of condition therapists are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem Solving Therapy as Usual (Active Comparator): Clinicians in this arm of care will have access to the Case Management Tracking System which is already in use.
  Intervention: unguided PST
  Interventions: Behavioral: Problem Solving Therapy as Usual
- Assisted Problem Solving Therapy (Experimental): This arm will be designed and finalized in Phase 1 and 2 of the project. We anticipate that the intervention will leverage clinical notes required to be completed by clinicians and will provide information to clinicians to help patients improve over time, as well as help clinicians implement PST to high quality.
  Intervention: guided PST
  Interventions: Behavioral: Assisted Problem Solving Therapy

INTERVENTIONS:
Behavioral: Problem Solving Therapy as Usual — Treatment as usual to deliver 6 weekly sessions to teach patients how to use the seven step process to solve problems.
  Other Names: Problem Solving Therapy
  Arms: Problem Solving Therapy as Usual
Behavioral: Assisted Problem Solving Therapy — Smart note assisted delivery of 6 weekly session to teach patients how to use the seven step process to solve problems
  Arms: Assisted Problem Solving Therapy

SUMMARY:
Problem Solving Therapy for Primary Care (PST-PC) is an evidence based psychosocial intervention (EBPI) for use in primary care settings, with more than 100 clinical trials.

Despite its proven efficacy we have found that implementation of PST-PC is complicated, resulting in rapid program drift (deviation from protocol with associated loss of efficacy), among practitioners following completion of training. Many studied have shown that program drift is not uncommon in the implementation of EBPIs and can be mitigated through on-going decision support and supervision. Unfortunately, decision support and supervisors of EBPIs are not widely available in low-resourced primary care clinics. We will address this problem by creating decision support tools to be integrated into electronic health records. Because these tools are deemed by many practitioners in other fields to be burdensome, we will explicitly involve active input on the content, design and function of these support tools. Outcomes may include electronic dashboards for panel management, automated suggestions for application of PST-PC elements based on patient reported outcomes or integration of automated patient tracking, and support of patient engagement. We hypothesize that enhanced decision support (target mechanism) will sustain quality delivery of PST-PC, which in turn will improve patient reported outcomes.

DETAILED DESCRIPTION:
Specific aims. Although evidence-based psychosocial interventions (EBPIs) are a preferred treatment option by vulnerable populations, they are rarely available in community primary care settings and when available, are often delivered with poor fidelity. High quality delivery of evidence-based psychosocial interventions (EBPIs) in primary care medicine is a function of many variables, including clinician training and usability of the intervention. Several studies find that for EBPIs to be delivered with sustained quality, on-going supervision and guidance is critical (this study's focus). While the availability of clinicians trained in EBPIs is scarce, the availability to supervisors trained in EBPIs is even more limited. Given the ubiquity of electronic health records, automated decision support tools and feedback systems have been found to be effective in supporting sustained quality EBPIs, but in practice have had mixed success on outcomes such that they may actually hinder clinical care and are often ignored by clinicians. In a report by the Agency for Healthcare Research and Quality, a significant barrier to the use of decision support tools is that these tools have not been developed with input from the clinician or in consideration of their work environment. Using the Center's Discover, Design, Build, Test (DDBT) framework, we will work with clinicians from 13 Behavioral Health Integration Program (BHIP) sites to create a clinical decision tool that addresses the common decisional dilemmas clinicians face when implementing EBPIs. We hypothesize that creating tools to support EBPIs will result in improved clinician competency and sustained skill (target) to EBPIs, compared to clinicians without these supports, resulting in better patient outcomes . The specific aims of this study are:

Aim 1: Discover Phase (6 months). Using Participant Action research (PAR) informed user-centered design methods we will interview clinicians in primary care about challenges they face in the delivery of two EBPIs, Behavioral Activation and Problem Solving Treatment, observe them delivering these EBPIs, and receiving feedback on cases from experts in these EBPIs. This process will help us to identify the common decisional dilemma's clinician's face in delivering EBPIs, their preferences for expert guidance strategies, and how decision support tools could be embedded into clinic workflow to reduce obstacles and enhance the delivery of EBPIs.

Aim 2: Design/Build Phase (6 months). Based on information obtained in the discover phase, we will engage in a rapid cycle iterative prototype development and testing of decision support tools to support PST-PC, to be carried out using user-centered design (UCD). The build of these tools will include the development of prototypes for user testing and refinement with input from care managers across the 13 BHIP sites. Data from this phase will be used to inform the Matrix of EBPI Modifications.

Aim 3: Test Phase (18 months) In the second to third year of the proposed project we will test the decision support tools in a small pilot trial with six providers and thirty patients randomized to the use of the decision support tools. H1: Clinicians with access to decision tools will report better acceptability, usability, and less burden when using PST-PC than clinicians without the tools. H2: Clinicians randomized to decision support tools will more competently deliver EBPI elements than clinicians randomized to unsupported EBPI. H3: Patients treated by clinicians with access to decision tools will have better patient-reported outcomes than patients treated by clinicians without access to these tools as assessed with functional disability and change in depression symptoms over time .

ELIGIBILITY:
Inclusion Criteria:

Clinicians: 18 years of age, able to read and speak English, provides psychotherapy as part of the University of Washington Medicine network, and willing to video-record PST sessions with patient participants Clients: 18+ years of age, able to read and speak English, willing to receive psychotherapy from a clinician who is also participating in the study, willing to have therapy sessions video-recorded, Patient Health Questionnaire-9 score of 10 or higher

Exclusion Criteria:

Client: History or presence of psychiatric diagnoses other than unipolar, non-psychotic depression or generalized anxiety disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Bennett, PhD, Study Chair — UWMC Psychiatry
Locations (1):
- Behavioral Health Integration Program, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Once data is collected and analyzed, we will make access to data available upon outreach to the principal investigator. Any interested party may have access to the data upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This data will be available by June 31, 2024 for up to five years.
Access Criteria: A request outlining the purpose of the data request, the length of time data will be stored before destruction, and the security protocol shall be sent to the study principal investigator for review.

REFERENCES:
- [Derived] Lyon AR, Munson SA, Renn BN, Atkins DC, Pullmann MD, Friedman E, Arean PA. Use of Human-Centered Design to Improve Implementation of Evidence-Based Psychotherapies in Low-Resource Communities: Protocol for Studies Applying a Framework to Assess Usability . JMIR Res Protoc. 2019 Oct 9;8(10):e14990. doi: 10.2196/14990. PMID 31599736

RESULTS

PARTICIPANT FLOW:
Groups:
- Problem Solving Therapy as Usual Clinicians: Clinicians in this arm of care had access to the Case Management Tracking System which is already in use.
  Intervention: unguided Problem Solving Therapy
  Problem Solving Therapy as Usual: Treatment as usual to deliver 6 weekly sessions to teach patients how to use the seven step process to solve problems.
- Assisted Problem Solving Therapy Clinicians: Clinicians in this arm of care had access to a Case Management and Problem Solving Therapy digitally assisted system
  Intervention: guided Problem Solving Therapy
  Assisted Problem Solving Therapy: Smart note assisted delivery of 6 weekly session to teach patients how to use the seven step process to solve problems
- Problem Solving Therapy as Usual Clients: Clients in this arm were served by clinicians in the Problem Solving Therapy as usual arm.
  Problem Solving Therapy as Usual: Treatment as usual to receive 6 weekly sessions to learn how to use the seven step process to solve problems.
- Assisted Problem Solving Therapy Clients: Clients in this arm were served by clinicians in the Problem Solving Therapy as usual arm.
  Assisted Problem Solving Therapy: Smart note assisted delivery of 6 weekly session to learn how to use the seven step process to solve problems
Period: Overall Study
Arm/Group | Problem Solving Therapy as Usual Clinicians | Assisted Problem Solving Therapy Clinicians | Problem Solving Therapy as Usual Clients | Assisted Problem Solving Therapy Clients
Started | 4 | 7 | 4 | 9
Completed | 2 | 5 | 4 | 9
Not Completed | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Problem Solving Therapy as Usual Clinicians | Assisted Problem Solving Therapy Clinicians | Problem Solving Therapy as Usual Clients | Assisted Problem Solving Therapy Clients | Total
Number analyzed (Participants) | 4 | 7 | 4 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (6.81) | 47.0 (15.1) | 56.5 (22.4) | 34.4 (10.6) | 41.9 (15.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Man | 0 | 3 | 2 | 2 | 7
  Gender: Woman | 4 | 4 | 2 | 6 | 16
  Gender: Agender | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 4 | 4 | 4 | 9 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 2 | 5 | 4 | 3 | 14
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 4 | 9 | 24
Patient Health Questionnaire [Mean (Standard Deviation); unit: score on a scale] — Population: Only clients completed outcome measures at baseline
  score on a scale
    number analyzed (Participants) | 0 | 0 | 4 | 9 | 13
    (all) |  |  | 17.25 (5.5) | 15.78 (4.68) | 16.23 (4.76)
Sheehan Disability Assessment Scale [Mean (Standard Deviation); unit: score on a scale] — Population: Only clients completed outcome measures at baseline.
  score on a scale
    number analyzed (Participants) | 0 | 0 | 4 | 9 | 13
    (all) |  |  | 17.25 (5.12) | 20.33 (5.12) | 19.38 (5.12)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention Measure
Description: The Acceptability of Intervention Measure is a four item measure of intervention acceptability, where each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable. Total scores depicted here are mean item scores and therefore the minimum and maximum values are 1 and 5. Higher scores mean more acceptable.
Time Frame: Clinicians: Six months after certification in the intervention. Clients: Six week follow-up
Population: All participants with baseline data
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Problem Solving Therapy as Usual Clients: Clients in this arm were served by clinicians in the PST as usual arm.
  Problem Solving Therapy as Usual: Treatment as usual to receive 6 weekly sessions to learn how to use the seven step process to solve problems.
- Assisted Problem Solving Therapy Clients: Clients in this arm were served by clinicians in the PST as usual arm.
  Assisted Problem Solving Therapy: Smart note assisted delivery of 6 weekly session to learn how to use the seven step process to solve problems
Arm/Group | Problem Solving Therapy as Usual Clinicians | Assisted Problem Solving Therapy Clinicians | Problem Solving Therapy as Usual Clients | Assisted Problem Solving Therapy Clients
Number analyzed (Participants) | 2 | 5 | 4 | 9
score on a scale | 4.13 (.53) | 4.25 (1.3) | 3.69 (1.03) | 4.31 (.43)
Statistical Analysis 1: Comparison: Problem Solving Therapy as Usual Clinicians vs Assisted Problem Solving Therapy Clinicians; Test type: Superiority — t-tests; p = 0.905, t-test, 2 sided
Statistical Analysis 2: Comparison: Problem Solving Therapy as Usual Clients vs Assisted Problem Solving Therapy Clients; Test type: Superiority — t-test; p = .320, t-test, 2 sided

2. Primary Outcome: User Burden Scale
Description: The User Burden Scale is a 20-item scale that assesses user burden when working with a system or technology. Each item is rated on a 0-4 scale, with a maximum score of 80 (high burden) and minimum score of 0 (low burden).
Time Frame: Clinicians: Six months follow-up after they have been certified in PST. Clients: six week follow-up timepoint
Population: All participants with follow-up timepoints
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Problem Solving Therapy as Usual Clinicians | Assisted Problem Solving Therapy Clinicians | Problem Solving Therapy as Usual Clients | Assisted Problem Solving Therapy Clients
Number analyzed (Participants) | 2 | 5 | 4 | 9
score on a scale | 13.5 (.71) | 5.8 (6.14) | 8.68 (8.94) | 8.53 (6.32)
Statistical Analysis 1: Comparison: Problem Solving Therapy as Usual Clinicians vs Assisted Problem Solving Therapy Clinicians; Test type: Superiority; p = .155, t-test, 2 sided — Not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Problem Solving Therapy as Usual Clients vs Assisted Problem Solving Therapy Clients; Test type: Superiority; p = .974, t-test, 2 sided — Not adjusted for multiple comparisons

3. Primary Outcome: System Usability Scale
Description: The System Usability Scale is a 10-item scale with each item ranked on a five point system of low to high usability. Items are ranked from 1=strongly disagree to 5=strongly agree. The scale score is calculated by adding the item scores and multiplying the total by 2.5, with 0 being the least and 100 being the maximum. A score of 68 or better is considered to be above average usability. As score less than 68 is considered to be poor usability. In this study, a score of 80 or more is considered our cut off for high usability.
Time Frame: Clinicians: 6 month follow-up after certification in PST. Clients: Six week follow-up
Population: All participants with follow-up data, and only those who experienced PST-Aid (therefore, "as usual" participants were not administered the measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Problem Solving Therapy as Usual Clinicians | Assisted Problem Solving Therapy Clinicians | Problem Solving Therapy as Usual Clients | Assisted Problem Solving Therapy Clients
Number analyzed (Participants) | 0 | 5 | 0 | 9
score on a scale |  | 75.5 (72.5) |  | 66.25 (68.8)

4. Secondary Outcome: Patient Health Questionnaire
Description: The Patient Health Questionnaire is a 9 item self report measure of depression, where each item is rated on a scale of 0-3, for a total possible score of 0-27. Higher scores are indicative of more depressed mood, with scores over 10 considered to be clinically depressed.
Time Frame: Baseline, 6 week follow-up
Population: Participants included all clients who reported data at follow-up. Clinicians did not complete this measure and therefore were not analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Problem Solving Therapy as Usual Clinicians | Assisted Problem Solving Therapy Clinicians | Problem Solving Therapy as Usual Clients | Assisted Problem Solving Therapy Clients
Number analyzed (Participants) | 0 | 0 | 4 | 9
score on a scale |  |  | 13.75 (2.99) | 10.33 (4.69)
Statistical Analysis 1: Comparison: Problem Solving Therapy as Usual Clients vs Assisted Problem Solving Therapy Clients; Test type: Superiority; p = .212, t-test, 2 sided

5. Secondary Outcome: Sheehan Disability Assessment Scale
Description: The Sheehan Disability Assessment Scale is 3-item self report measure of functioning, where each item is ranked on a scale of 1-10, with 1 = no disability and 10 =high disability, for a total scale score ranging from 0 to 30. Higher scores reflect greater disability.
Time Frame: Baseline, 6 week follow up
Population: Analysis on all clients who completed measures at 6 week follow-up. Clinicians did not complete this measure and are not analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Problem Solving Therapy as Usual Clinicians | Assisted Problem Solving Therapy Clinicians | Problem Solving Therapy as Usual Clients | Assisted Problem Solving Therapy Clients
Number analyzed (Participants) | 0 | 0 | 4 | 9
score on a scale |  |  | 15.25 (4.86) | 17.89 (6.90)
Statistical Analysis 1: Comparison: Problem Solving Therapy as Usual Clients vs Assisted Problem Solving Therapy Clients; Test type: Superiority; p = .507, t-test, 2 sided

6. Secondary Outcome: Problem Solving Therapy Clinician Certification
Description: Problem Solving Therapy Clinician Certification was determined using the Problem Solving Therapy Adherence Scale, an observer-rated, 11 item scale, with each scale raking therapist competency in delivering the seen steps of PST using a 0 (not competent) to 5 (expert level) scale. Coders then use these item scores to rate a global fidelity rating on the same 0 to 5 scale. Receiving a 3 or higher on two sessions resulted in certification to practice PST. Therefore the outcome of importance is a dichotomous "certified/not certified". We report here on the number of clinicians in each group who certified.
Time Frame: Expert clinicians reviewed audiotapes of therapy sessions for each clinician participant over a six month period of time after initial training.
Population: Therapists who submitted audiotapes for review by expert coders. PST adherence was not conducted for clients.
Measure: Count of Participants; unit: Participants
Arm/Group | Problem Solving Therapy as Usual Clinicians | Assisted Problem Solving Therapy Clinicians | Problem Solving Therapy as Usual Clients | Assisted Problem Solving Therapy Clients
Number analyzed (Participants) | 3 | 5 | 0 | 0
Participants | 1 | 5 |  |
Statistical Analysis 1: Comparison: Problem Solving Therapy as Usual Clinicians vs Assisted Problem Solving Therapy Clinicians; Test type: Superiority; p = .091, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Clinicians: 7 months. Clients: 6 weeks.
Arm/Group | Problem Solving Therapy as Usual Clinicians | Assisted Problem Solving Therapy Clinicians | Problem Solving Therapy as Usual Clients | Assisted Problem Solving Therapy Clients
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/4 | 0/9
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/4 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT03516513/Prot_SAP_000.pdf